CLINICAL TRIAL: NCT00004244
Title: Phase I Trial of rhIL-12 and rHuIFN-a2b in Patients With Metastatic Renal Cell Carcinoma or Malignant Melanoma
Brief Title: Interleukin-12 and Interferon Alfa in Treating Patients With Metastatic Kidney Cancer or Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067489; CCF-IRB-3063; NCI-T99-0028
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2005-06

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — Interferon-alpha; Interleukin-12 Subunit p35

ARMS (3):
- Arm I (Experimental): Patients receive interleukin-12 subcutaneously (SC) twice a week and interferon alfa SC three times a week every week for 4 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression.
  Cohorts of 3-6 patients receive escalating doses of interleukin-12 and interferon alfa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.
  Patients receive interleukin-12 SC twice a week for 2 weeks, followed by treatment with interleukin-12 in combination with interferon alfa as described above.
  Interventions: Biological: recombinant interferon alfa; Biological: recombinant interleukin-12
- Arm II (Experimental): Patients receive interleukin-12 subcutaneously (SC) twice a week and interferon alfa SC three times a week every week for 4 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression.
  Cohorts of 3-6 patients receive escalating doses of interleukin-12 and interferon alfa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.
  Patients receive interferon alfa SC three times a week for 2 weeks, followed by treatment with interleukin-12 in combination with interferon alfa as described above.
  Interventions: Biological: recombinant interferon alfa; Biological: recombinant interleukin-12
- Arm III (Experimental): Patients receive interleukin-12 subcutaneously (SC) twice a week and interferon alfa SC three times a week every week for 4 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression.
  Cohorts of 3-6 patients receive escalating doses of interleukin-12 and interferon alfa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.
  Patients receive treatment with interleukin-12 in combination with interferon alfa at the MTD as described above.
  Interventions: Biological: recombinant interferon alfa; Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: recombinant interleukin-12

SUMMARY:
This phase I trial is studying the side effects and best dose of interleukin-12 and interferon alfa in treating patients with metastatic kidney cancer or malignant melanoma. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells. Interferon alfa may interfere with the growth of cancer cells. Combining interleukin-12 and interferon alfa may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity of interleukin-12 and interferon alfa in patients with metastatic renal cell carcinoma or malignant melanoma.

II. Determine the maximum tolerated dose of these drugs when concurrently administered in this patient population.

III. Obtain preliminary data on the antitumor efficacy of this combination in these patients.

OUTLINE: This is a dose-escalation study, followed by a randomized study.

Patients receive interleukin-12 subcutaneously (SC) twice a week and interferon alfa SC three times a week every week for 4 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of interleukin-12 and interferon alfa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.

Once the MTD is established, additional patients are accrued and randomized to 1 of the following treatment arms:

ARM I: Patients receive interleukin-12 SC twice a week for 2 weeks, followed by treatment with interleukin-12 in combination with interferon alfa as described above.

ARM II: Patients receive interferon alfa SC three times a week for 2 weeks, followed by treatment with interleukin-12 in combination with interferon alfa as described above.

ARM III: Patients receive treatment with interleukin-12 in combination with interferon alfa at the MTD as described above.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for the dose escalation portion of this study. An additional 18 patients (5 in arm I, 5 in arm II, and 8 in arm III) will be accrued to the randomized portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma or malignant melanoma
* Strong clinical evidence or biopsy proof of metastases to a site or sites distant from the primary tumor
* Bidimensionally measurable of evaluable disease
* No significant effusions and/or ascites
* No more than 3 prior regimens for metastatic disease
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.5 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* ALT/AST no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 1.8 mg/dL
* Calcium no greater than 11.5 mg/dL

Cardiovascular:

* No history of serious cardiac arrhythmia or cardiac arrhythmia requiring treatment
* No congestive heart failure
* No angina pectoris
* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active peptic ulcer
* No autoimmune disease
* No inflammatory bowel disease
* No local or systemic infections requiring IV antibiotics within the past 28 days
* No known seizure disorder
* No other prior malignancy except basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any curatively treated malignancy in complete remission for at least 3 years
* HIV, hepatitis B surface antigen, and hepatitis C negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior biologic therapy

Chemotherapy:

* Recovered from prior chemotherapy

Endocrine therapy:

* At least 28 days since prior hormonal therapy and recovered
* No concurrent corticosteroids except for replacement steroids

Radiotherapy:

* Recovered from prior radiotherapy
* At least 28 days since prior radiotherapy for control of pain from skeletal lesions

Surgery:

* At least 28 days since prior major surgery requiring general anesthesia
* No organ allografts

Other:

* No concurrent aspirin
* No concurrent barbiturates
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-03; Primary Completion 2005-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M. Bukowski, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States